CLINICAL TRIAL: NCT06809543
Title: Clinical Benefits and Safety of Tropho Tend in the Management of Painful Rotator Cuff Tendinopathy (RCT)
Brief Title: Clinical Benefits and Safety of Tropho Tend in the Management of Painful Rotator Cuff Tendinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mastelli S.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tropho-Try-2024
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Tendinopathy
Keywords: Polynucleotides; PN HPT; Mastelli; Rotator cuff tendinopathy; Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy group (Experimental)
  Interventions: Device: Polynucleotides (Tropho Tend)
- Control group (Active Comparator)
  Interventions: Procedure: Rehabilitation physiotherapy

INTERVENTIONS:
Device: Polynucleotides (Tropho Tend) — Tropho Tend is administered by injecting the solution at level of muscular-tendineal (MJT) or osteo-tendineal junctions (OTJ) using a fine-gauge needle (usually 25-30G).
  Before injecting the product, the target area will be disinfected with alcohol or another antiseptic, with the antiseptic removed with physiologic sterile solution.
  Total number of treatments will consist in 3 Tropho Tend administrations: at T0 - basal visit;
  * T1 - after 2 weeks;
  * T3 - after 4 weeks.
  Arms: Therapy group
Procedure: Rehabilitation physiotherapy — Rehabilitation physiotherapy (standard of care)
  Arms: Control group

SUMMARY:
This is a prospective, open label, controlled, exploratory clinical investigation aimed to evaluate the clinical benefit and safety of Tropho Tend in the conservative management of painful Rotator Cuff Tendinopathy (RCT).

All subjects will be involved in the clinical investigation for 4 months for a total of 5 visits (T0= basal visit, T1, T2, T3, T4).

The control group will be represented by patients diagnosed with rotator cuff tendinopathy treated with rehabilitation physiotherapy (standard of care).

The therapy group will be represented by patients diagnosed with rotator cuff tendinopathy treated with rehabilitation physiotherapy + TrophoTend perilesional injection (TrophoTend will be added on to current standard of care).

All the screened patients at the baseline visit (T0), after checking the inclusion/exclusion criteria, will be prospectively included in the clinical investigation, in a 1:1 randomization. Patients will be randomly assigned to the "control group" (N=30pts), receiving rehabilitation physiotherapy (standard of care), or to the "therapy group" (N=30 pts), receiving Tropho Tend as a add on therapy to the rehabilitation physiotherapy.

Total duration of Clinical Investigation will be 12 months: 2-4 months for patients screening and enrolment; 1 month of therapy administration (3 perilesional injections 2 weeks apart); 3 months of follow-up; 2-4 months for data analysis and final report/paper elaboration.

At the baseline visit (T0), an ultrasound evaluation (EUS) has to be performed to assess tendon condition. If an EUS evaluation performed within one month from T0 is available, this will be considered acceptable. This first evaluation has to be compared with another EUS performed at the final visit to obtain a qualitative description of the ultrasound appearance of the tendon after the treatment.

Patients' enrolment will take 2-4 months. Tropho Tend will be administrated at T0 (basal visit) at T1 (2 weeks) and at T2 (4 weeks) for a total duration of treatment of 1 month.

Follow-up will be performed at T3 (8 weeks) and T4 (12 weeks= 3 months). End of the clinical investigation will be considered the last visit for the last enrolled patient.

A 40% reduction in mean VAS scores between the "Tropho Tend therapy group" and the "control group" is considered as reflecting meaningful clinical improvement for the patient.

At the final visit, the patient has to rate his/her satisfaction with the treatment using a 5-points Likert scale, where 1=very dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied, 5=highly satisfied.

ELIGIBILITY:
Inclusion Criteria

* Male and female patients ≥ 18 years of age, in good general health condition.
* Painful Rotator Cuff Tendinopathy (RCT) since ≥ 6 weeks.
* Pain and impaired functionality on a 0 to 10 cm-centimeter specifically designed Visual Analogue Scale (VAS) ≥ 4 cm at baseline visit.
* Rotator Cuff Tendinopathy (RCT) diagnosis, based on clinical examination.
* Tendon ultrasound (EUS) performed within one month of enrollment.
* Signed written informed consent.

Exclusion Criteria

* Treatment with any investigational product within 6 months prior to clinical investigation entry.
* Patients with known hypersensitivity to the products (active compound and excipients) or any component or procedure used in the clinical investigation.
* Patients with para-tendinopathy, partial/total rupture, previous tendon surgery.
* Severe intercurrent illness (e.g.: uncontrolled diabetes mellitus, peripheral neuropathy, autoimmune or inflammatory condition, metabolic disorders, severe oncological conditions) that, in the opinion of the investigator, may put the patient at risk when participating in the clinical investigation or affect the patient's ability to take part in the clinical investigation .
* Patients treated with systemic and/or local steroids within the last 6 months, immunosuppressive drugs within the last 3 months, repeated use of non-steroidal anti-inflammatory drugs (NSAIDs) within the last week or occasional use within 24 hours.
* Recent history of drug and/or alcohol abuse (within the last 6 months).
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Variation of pain and functional impairment | All visits from baseline to the last follow-up after 12 weeks from the end of the treatment
  The Primary Endpoint measure is the variation of VAS Visual Analogue Scale of pain and of function (VAS; 0-10 cm, where 0= no pain or no function impairment and 10= worse pain or function impairment) in the "Tropho Tend therapy group" compared with the "control group". A 40% reduction in mean VAS scores between the "Tropho Tend therapy group" and the "control group" is considered as reflecting meaningful clinical improvement for the patient.
Variation of Shoulder pain and disability index (SPADI) between the 2 groups | All visits from baseline to the last follow-up after 12 weeks from the end of the treatment
  SPADI Index is designed to measure current shoulder pain and function of daily tasks in an outpatient setting.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.
  The pain dimension consists of five questions regarding the severity of an individual's pain.
  Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
Single assessment numeric evaluation (SANE) | All visits from baseline to the last follow-up after 12 weeks from the end of the treatment
  The Primary Endpoint measure is also the change from baseline of the single assessment numeric evaluation (SANE), which was designed as a simple one-question: "how would you rate your shoulder today as a percentage of normal (0% to 100%, with 100% being normal)?"

SECONDARY OUTCOMES:
Patient's satisfaction | From the second visit (T1) to last follow-up after 12 weeks from end of treatment
  Patient's satisfaction with the treatment using a 5-points Likert scale (1=very dissatisfied, 2=dissatisfied, 4=neutral, 4=satisfied, 5=highly satisfied). A final score of 2 points or more on the Likert scale at the last clinical investigation visit will be considered clinically significant.
Qualitative description of the ultrasound appearance of the tendon | Baseline and last follow-up visit (T4)
  A qualitative description of the ultrasound appearance of the tendon will be required to compare the final follow-up visit to that of an ultrasound performed at the baseline visit in both groups
Quality of Life using EQ-5D-3L Paper Self-Complete | Baseline and at the two follow-up visits (at T3 - 8 weeks after the end of the treatment and T4 - 12 weeks after the end of the treatment)
  The EQ-5D-3L descriptive system comprises the following five dimensions, each describing a different aspect of health: MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems. The respondent is asked to indicate his / her health state by checking the box against the most appropriate statement in each of the five dimensions. The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents. The scale used for the answers is the EQ visual analogue scale (EQ VAS). It consists of a vertical 100 point visual analogue scale with two extreme endpoints (0= worst health status; 100=best health status).
Adverse events (AE) monitoring | All visits from baseline to the last follow-up after 12 weeks from the end of the treatment
  Adverse events (AE) will be monitored throughout the trial. At each scheduled visit, a safety assessment has to be conducted by the investigator. The intensity (mild/moderate/severe) will be assessed according to the investigator's judgement. If a patient drops out of the clinical investigation, the possible reasons for drop-out, including no improvement in the tendinopathy or occurrence of unacceptable signs/symptoms, need to be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Sassuolo S.p.A., Sassuolo, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Colangelo MT, Govoni P, Belletti S, Squadrito F, Guizzardi S, Galli C. Polynucleotide biogel enhances tissue repair, matrix deposition and organization. J Biol Regul Homeost Agents. 2021 Jan-Feb;35(1):355-362. doi: 10.23812/20-320-L. No abstract available. PMID 33480222
- [Result] Saggini R, Khodor HH, Capogrosso F, Carniel R, Bellomo RG. La condro-sincronizzazione nel danno articolare complesso: risultati della viscosupplementazione con Condrotide. Journal of viscosupplementation.it 2016; 2(1): 1-7.
- [Result] Saggini R, Di Stefano A, Capogrosso F, Carniel R, Haidar Hassan K, et al. (2014) Viscosupplementation with Hyaluronic Acid or Polynucleotides: Results and Hypothesis for Condro-synchronization. J Clin Trials 4: 198. doi:10.4172/2167-0870.1000198